CLINICAL TRIAL: NCT01898182
Title: A Single Arm, Phase IV, Open-Label, Split-Face Trial to Evaluate the Efficacy and Safety of Kinetin, N6-furfuryladenine, 0.1% for Treatment of Cutaneous Photoaging
Brief Title: Efficacy and Safety of Kinetin 0.1% for Treatment of Skin Photoaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makati Medical Center (Other)
Collaborators: A. Menarini Philippines, Inc. (Industry)
Responsible Party: Principal Investigator, Ma. Purita Paz-Lao, MD, FPDS, Chairman, Makati Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MMCDeptofDerma-Kinerase-2013
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Cutaneous Photoaging
MeSH Terms: interventions — Kinetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kinerase (Experimental): Kinetin (N6-furfuryladenine) is an essential bio growth factor that regulates cell growth and is proven to delay and reverse the signs of aging. Kinerase has been found out to significantly improve the appearance of skin texture, mottled hyperpigmentation and fine wrinkles. It does not cause the cutaneous side effects that result from other commonly used anti-aging products. The Kinerase cream contains: Water, glyceryl stearate, propylene glycol, butylenes glycol, glycerin, cetyl alcohol, stearic acid, isopropyl palmitate, squalene, stearyl alcohol, glycene soja sterols, dimethicone, laureth-23, aloe barbadensis leaf juice, phenoxyethanol, carbomer, ethylhexyglycerin, sodium hydroxide, soluble collagen, kinetin, panthenol, tocopherol, citric acid, sodium citrate, hydrolysed elastin.
  Interventions: Other: Kinetin, N6-furfuryladenine, 0.1%

INTERVENTIONS:
Other: Kinetin, N6-furfuryladenine, 0.1%
  Other Names: Kinerase cream

SUMMARY:
The purpose of the study is to evaluate the change in the severity and clinical signs of skin photoaging among Filipino patients using Kinerase cream (Kinetin 0.1%). This study will recruit 132 subjects from dermatological clinics in a tertiary hospital in the Philippines for a period of 3 months (12 weeks). Changes in severity will be documented using physician evaluation, self-evaluation, and through VISIA complexion analysis system.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, split-face trial in subjects with mild to moderate photoaged facial skin. The study will enroll around 132 subjects from selected private dermatology clinics in a tertiary hospital in the Philippines.

Patients from selected private dermatology clinics of a tertiary hospital will be screened and recruited to participate. They will be provided a written consent form (Appendix I) before they will be included in the study.

Following enrollment, subjects will return for outpatient visits at weeks 4, 8, and 12 for assessment.

The whole study will be conducted from July 2013 to November 2013. The first month would involve recruitment of patients. Qualified patients will start the 12-week treatment period and will be asked to follow up every 4 weeks. The last two months would be for data analysis, interpretation and writing of the scientific report.

ELIGIBILITY:
Inclusion Criteria:

* Filipino and Asian female subjects from private clinics of a tertiary hospital in the Philippines older than 35 years of age and less than 65 years of age.
* Subjects with mild to moderate cutaneous photoaging as assessed by the investigator's assessment 6-point scale.
* Subjects willing to sign an informed consent and adhere to all protocol requirements.

Exclusion Criteria:

* Suspected porphyria, systemic or cutaneous lupus erythematosus, or any other photosensitizing disorder or drug-induced photosensitization
* Chronic or recurring skin disease or disorder
* Any active infectious skin disorder (Herpes simplex, molluscum contagiosum, and facial warts)
* Skin cancer of the facial tissues
* Any laser/IPL/ chemical peel in the 2 months preceding the screening visit
* History of Isotretinoin use, 6 months prior to the screening disease
* Topical tretinoin or adapalene in the 2 months prior to the screening visit
* Used topical alpha-hydroxy acid skincare products in the month preceding the screening visit
* On any anti-aging products and who wish to continue use of their products
* Requiring concurrent treatment that would interfere with the study assessments
* Pregnant or lactating females

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Skin Roughness | 12 weeks
  Measured using Physician Evaluation and Patient Self-Evaluation of severity of cutaneous photoaging at baseline week, weeks 4, 8, and 12
Pigmentation | 12 weeks
  Also called Mottling or Blotchiness. This is measured using Physician Evaluation and Patient Self-Evaluation of severity of cutaneous photoaging at baseline week, weeks 4, 8, and 12
Fine wrinkles | 12 weeks
  Measured using Physician Evaluation and Patient Self-Evaluation of severity of cutaneous photoaging at baseline week, weeks 4, 8, and 12
Global Improvement in Cutaneous Photoaging | 12 weeks
  Measured using Physician Evaluation and Patient Self-Evaluation of severity of cutaneous photoaging at baseline week, weeks 4, 8, and 12
Pores | 12 weeks
  Measured using VISIA Complexion Analysis System at baseline week, weeks 4 and 8.
Wrinkles | 12 weeks
  Measured using VISIA Complexion Analysis System at baseline week, weeks 4 and 8.
Texture | 12 weeks
  Measured using VISIA Complexion Analysis System at baseline week, weeks 4 and 8.
Porphyrins | 12 weeks
  Measured using VISIA Complexion Analysis System at baseline week, weeks 4 and 8.
Visual Spots | 12 weeks
  Measured using VISIA Complexion Analysis System at baseline week, weeks 4 and 8.
UV spots | 12 weeks
  Measured using VISIA Complexion Analysis System at baseline week, weeks 4 and 8.
Brown Spots | 12 weeks
  Measured using VISIA Complexion Analysis System at baseline week, weeks 4 and 8.
Red Areas | 12 weeks
  Measured using VISIA Complexion Analysis System at baseline week, weeks 4 and 8.

SECONDARY OUTCOMES:
Erythema | 12 weeks
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a test product and which does not necessarily have a casual relationship with this treatment (ICH-GCP definition). In this study, all untoward medical occurrences will be collected irrespective whether the subject has taken any study product or not.
Burning | 12 weeks
  Also includes stinging. An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a test product and which does not necessarily have a casual relationship with this treatment (ICH-GCP definition). In this study, all untoward medical occurrences will be collected irrespective whether the subject has taken any study product or not.
Peeling | 12 weeks
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a test product and which does not necessarily have a casual relationship with this treatment (ICH-GCP definition). In this study, all untoward medical occurrences will be collected irrespective whether the subject has taken any study product or not.
Pruritus | 12 weeks
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a test product and which does not necessarily have a casual relationship with this treatment (ICH-GCP definition). In this study, all untoward medical occurrences will be collected irrespective whether the subject has taken any study product or not.
Dryness | 12 weeks
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a test product and which does not necessarily have a casual relationship with this treatment (ICH-GCP definition). In this study, all untoward medical occurrences will be collected irrespective whether the subject has taken any study product or not.
Edema | 12 weeks
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a test product and which does not necessarily have a casual relationship with this treatment (ICH-GCP definition). In this study, all untoward medical occurrences will be collected irrespective whether the subject has taken any study product or not.
Acne | 12 weeks
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a test product and which does not necessarily have a casual relationship with this treatment (ICH-GCP definition). In this study, all untoward medical occurrences will be collected irrespective whether the subject has taken any study product or not.

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Purita P. Lao, MD, FPDS, Principal Investigator — Makati Medical Center
Locations (2):
- Philippines (2):
  - Makati Medical Center, Makati City, National Capital Region
  - Makati Medical Center Department of Dermatology, Makati City, NCR